CLINICAL TRIAL: NCT04990661
Title: The Effect of the Massage on Cramp Frequency, Cramp Severity, and Sleep Quality of Hemodialysis Patients With Complaint of Cramp
Brief Title: The Effect of the Massage on Cramp Frequency, Cramp Severity, and Sleep Quality
Acronym: Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Ayse Gul Parlak, Lecturer, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kafkas Unıversity
Record Dates: First submitted 2021-07-02; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Muscular Cramps; Hemodialysis
Keywords: Hemodialysis; massage; muscle cramps; sleep quality
MeSH Terms: conditions — Muscle Cramp; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (massage group) (Experimental): intradialytic massage for lower extremity was applied to the intervention group in three sessions a week and a total of six sessions for two weeks
  Interventions: Behavioral: intradialytic massage
- Control group (No Intervention): not administered except nursing interventions in the HD unit.

INTERVENTIONS:
Behavioral: intradialytic massage — intradialytic massage for lower extremity ( the massage included both feet and legs up to and including the knee) applied to the intervention group in three sessions a week and a total of six sessions for two weeks
  Arms: Intervention group (massage group)

SUMMARY:
The aim of this randomized controlled experimental study was to determine the effect of the massage applied to hemodialysis patients with complaint of cramp on the cramp frequency, cramp severity, and sleep quality.

DETAILED DESCRIPTION:
The study was conducted with patients receiving treatment in a total of four hemodialysis units. The sample of the study comprised a total of 36 patients (18 patients in the intervention group and 18 patients in the control group) with complaint of cramp. In the study, intradialytic massage for lower extremity was applied to the intervention group in three sessions a week and a total of six sessions for two weeks. No intervention other than routine care was applied to the control group patients.

In the study, the data were collected using a patient information form, cramp assessment short survey, the "Visual Analog Scale (VAS)", "Pittsburgh Sleep Quality Index" (PUKİ), and patient follow-up forms.

In order to conduct the study, the necessary Ethics Committee approval and institutional permission were obtained. The individuals included in the study informed about the purpose of the research, their verbal consent obtained and the participant's informed consent form signed.

After the intervention and control groups were assigned according to the research criteria, the days and sessions of the groups were determined and recorded in the digital randomization environment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years,
* One or more lower work cramp attacks during/after dialysis
* Have a constant dryness in the last 1 month (few changes weighing more than 2 kg)
* Receiving at least 6 hemodialysis treatments
* Receiving hemodialysis treatment 3 times a week
* Those who have not received sub-massage therapy before

Exclusion Criteria:

* Having one of the diagnoses of chronic obstructive pulmonary disease, cancer, psychiatric disease
* Presence of any soft tissue, nerve and vascular disease in the lower extremities
* Presence of infection, open wound, suspected fracture, dermatitis, burn and edema in the lower extremities
* Having had a lower extremity operation in the past six weeks
* Receiving hemodialysis treatment for less than 6 months (new patients are excluded because the first few months of dialysis treatment are periods of hemodynamic instability)
* Having a fluctuating dry weight (excluded from the study as it may cause cramping)
* Having been diagnosed with neuropathy in the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala (VAS) | during 2 weeks (15 days)
  This scale; There is a number value of "0 (no pain)" at the beginning and "10 (the most unbearable pain)" at the end. Participants marked the scale each time they experience a muscle cramp severity. Baseline measurements; muscle cramp experienced at home and, during the dialysis session.
Muscle cramp assessment short survey (duration and frequency of muscle cramps) | during 2 weeks (15 days)
  Participants noted the duration and number of muscle cramps they experienced. Baseline measurements; muscle cramp experienced at home and, during the dialysis session.
Patient follow-up forms. | during 2 weeks (15 days)
  Intradialytic systolic and diastolic blood pressure and ultrafiltration were noted by the investigator, during the HD session

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index(PUKİ), | At the first and last meeting in 2 weeks (15 days)
  Pittsburgh Sleep Quality Index (PUKI) used to evaluate sleep quality.The total score is between 0-21. PUKİ score of 5 or above indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: ayşe gül parlak, Principal Investigator — Kafkas Üniversity
Locations (2):
- Turkey (Türkiye) (2):
  - Ayşe Gül Parlak, Kars
  - Kafkas University, Kars

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mastnardo D, Lewis JM, Hall K, Sullivan CM, Cain K, Theurer J, Huml A, Sehgal AR. Intradialytic Massage for Leg Cramps Among Hemodialysis Patients: a Pilot Randomized Controlled Trial. Int J Ther Massage Bodywork. 2016 Jun 3;9(2):3-8. doi: 10.3822/ijtmb.v9i2.305. eCollection 2016 Jun. PMID 27257445
- [Background] Cox KJ, Parshall MB, Hernandez SHA, Parvez SZ, Unruh ML. Symptoms among patients receiving in-center hemodialysis: A qualitative study. Hemodial Int. 2017 Oct;21(4):524-533. doi: 10.1111/hdi.12521. Epub 2016 Dec 19. PMID 27990732
- [Background] Flythe JE, Hilliard T, Lumby E, Castillo G, Orazi J, Abdel-Rahman EM, Pai AB, Rivara MB, St Peter WL, Weisbord SD, Wilkie CM, Mehrotra R; Kidney Health Initiative Prioritizing Symptoms of ESRD Patients for Developing Therapeutic Interventions Stakeholder Meeting Participants. Fostering Innovation in Symptom Management among Hemodialysis Patients: Paths Forward for Insomnia, Muscle Cramps, and Fatigue. Clin J Am Soc Nephrol. 2019 Jan 7;14(1):150-160. doi: 10.2215/CJN.07670618. Epub 2018 Nov 5. PMID 30397026